CLINICAL TRIAL: NCT04441450
Title: Absorption, Metabolism, and Excretion of Oral 14C Radiolabeled ICP-022: An Open-Label, Phase I, Single-Dose Study in Healthy Males
Brief Title: ADME Study of [14C]ICP-022 in Healthy Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICP-CL-00110
Record Dates: First submitted 2020-06-16; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]ICP-022 (Experimental): Subjects will take a single of 150mg 100μCi of [14C]ICP-022.
  Interventions: Drug: [14C]ICP-022

INTERVENTIONS:
Drug: [14C]ICP-022 — 150mg suspension containing 100μCi of [14C]ICP-022

SUMMARY:
The purpose of this study is to investigate the absorption, the metabolic pathways and the excretion of ICP-022 in healthy male adult participants after administration of a single oral dose of 150 mg of 14C ICP-022.

ELIGIBILITY:
key Inclusion criteria:

1. Weight: Body mass index (BMI) is 19~26 kg/m2
2. signing of informed consent
3. Volunteers are able to communicate well with the investigators and be able to complete the trial according to the process

Key Exclusion Criteria:

1. physical examination, vital signs, routine laboratory tests (blood routine, blood biochemistry, blood coagulation routine, urine routine, stool routine + occult blood, serum amylase, thyroid function, etc.), 12-lead ECG, Chest X-ray (Anteroposterior), abdominal B-ultrasound (hepatobiliary, pancreas, spleen and kidney) and other abnormalities and clinical significance.
2. ophthalmologic examination shows abnormality and clinical significance
3. Positive test for hepatitis B (surface antigens HBs), or C (antibody HCs), positive test for HIV, positive test for Syphilis antibody.
4. Within 1 month before the screening, having not limited to known as hepatic enzyme inducers, inhibitors or substrates; (eg, inducer - barbiturate, carbamazepine, phenytoin, rifampicin, dexamethasone, rifabutin, rifapentine; inhibitors - SSRI antidepressants, cimetidine, diltiazem, macrolides, verapamil, imidazole antifungals) ;
5. Within 1 month before the screening, receiving the anticoagulant therapy such as warfarin or thrombin inhibitor and/or aspirin antiplatelet therapy

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Distribution ratio of total radioactivity in whole blood and plasma of [14C]ICP-022 | Up to14 days
  To investigate the pharmacokinetics of total radioactivity in plasma after oral [14C] ICP-022 in healthy volunteers, and the distribution ratio of total radioactivity in whole blood and plasma.
Quantitative analysis of total radioactivity in excreta after oral [14C] ICP-022 in healthy volunteers | Up to14 days
  Quantitative analysis of total radioactivity in excreta after oral [14C] ICP-022 in healthy volunteers, obtaining body material balance data and main excretion pathways

SECONDARY OUTCOMES:
Quantitative analysis of the concentration of ICP-022 in plasma | Up to14 days
  Quantitative analysis of the concentration of ICP-022 in plasma to obtain the pharmacokinetic parameters of ICP-022
The biotransformation pathways of [14C]ICP-022 | Up to14 days
  Urine and fecal collection for metabolite profiling. Identify the main metabolites in humans after oral [14]ICP-022 in healthy volunteers to determine the main biotransformation pathways.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No